CLINICAL TRIAL: NCT03762837
Title: Multicenter Prospective Cohort Study of Risk Factors for Gallbladder Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TJ-IRB20181109
Record Dates: First submitted 2018-12-02; First posted 2018-12-04 (Actual); Last update posted 2019-03-04 (Actual); Status verified 2018-11

CONDITIONS: Gallbladder Diseases; Healthy
Keywords: Gallbladder cancer
MeSH Terms: conditions — Gallbladder Diseases; Gallbladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposure group：Benign gallbladder disease: Patients with benign gallbladder diseases, such as gallbladder polyps, gallstones, etc.
  Interventions: Other: Benigh gallbladder diseases
- Non-exposed group: healthy people: Patients without benign gallbladder diseases

INTERVENTIONS:
Other: Benigh gallbladder diseases — We aim to observe the relationship between the benigh gallbladder diseases and gallbladder cancer, and we will not take any actions to interrupt.
  Groups: Exposure group：Benign gallbladder disease

SUMMARY:
This trial is a prospective study, the main purpose of the study is to investigate the association between benign gallbladder disease and gallbladder carcinoma; to explain the timing of intervention, intervention and early prevention of benign gallbladder disease; according to the national epidemiology of gallbladder cancer Center Clinical Research (unpublished), 2000 National Cholecystoma Clinical Epidemiology Report, and 2005 Clinical Analysis of 2379 Cases of Gallbladder Carcinoma in 17 Hospitals in Five Northwest Provinces, Pre-experimental data, using samples The volume estimation formula, α = 0.05, β = 0.1, plans to enroll 100,000 people.Half of participants is someone with Biliary benign disease，while the other half is healthy.

DETAILED DESCRIPTION:
Gallbladder cancer is the most common malignant biliary tract tumor. The main risk factors for gallbladder cancer include gallstones, gallbladder polyps, gallbladder adenomas, chronic inflammation of the gallbladder, etc. However, recently, there is still a lack of evaluation data on relevant risk factors. Therefore, on the basis of large-scale epidemiological investigations, large-scale prospective studies are needed to further clarify the level of risk factors associated with gallbladder cancer. With the development of modern imaging technology and deep understanding of gallbladder diseases, the detection rate of benign gallbladder lesions (cacerous polyps, gallbladder adenomyosis, gallbladder adenoma, gallstones, etc.) has increased year by year, and some benign gallbladder lesions can pass A series of pathophysiological processes have gradually evolved into gallbladder cancer. This study aimed to establish a prospective cohort of benign gallbladder disease, to explore the correlation, intervention time and socioeconomic benefits of benign gallbladder disease and gallbladder cancer. In order to further understand the current trend and diagnosis and treatment of benign gallbladder disease in China, the Chinese Society of Surgery Branch of the Chinese Society of Surgery will launch a national epidemiological survey of gallbladder cancer (2018). This study will provide a more detailed basis for the diagnosis and treatment of benign gallbladder disease in China.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who met the following four criteria entered the study.

  1. A benign gallbladder disease is detected during a medical examination or visit (according to any imaging test);
  2. healthy people without gallbladder disease;
  3. Age greater than 18 years and less than 80 years old;
  4. Sign the informed consent form. PS: If someone meets the condition (1) or (2), then he can be enrolled.

Exclusion Criteria:

* Subjects can not enter the study by combining any of the following

  1. Concomitant diseases such as severe mental illness, severe heart, lung and kidney;
  2. Refusal of follow-up requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The recruits included patients with benign gallbladder cancer and healthy people, mainly from the Grade-A Tertiary Hospitals and medical centers in China.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Gallbladder cancer | 3 years
  Comparison of incidence of gallbladder cancer between the two groups

DOCUMENTS (2):
  • Informed Consent Form (2018-08-31): https://cdn.clinicaltrials.gov/large-docs/37/NCT03762837/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2018-08-31): https://cdn.clinicaltrials.gov/large-docs/37/NCT03762837/Prot_SAP_001.pdf